CLINICAL TRIAL: NCT06788002
Title: Low-dose Radiotherapy and Chemoimmunotherapy in Nasopharyngeal Carcinoma With Liver Metastasis
Brief Title: LDRT and Chemoimmunotherapy in NPC With Liver Metastasis
Acronym: Light
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, HuaiLiu, Professor, Hunan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024528; Z2023080 (Other Grant/Funding Number: Hunan Provincial Health Commission)
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: nasopharyngeal carcinoma; liver metastasis; low-dose radiotherapy; chemotherapy; immunotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LDRT and chemoimmunotherapy (Experimental): Low-dose radiotherapy, chemotherapy, immunotherapy
  Interventions: Other: Low-dose radiotherapy combine with chemoimmunotherapy

INTERVENTIONS:
Other: Low-dose radiotherapy combine with chemoimmunotherapy — Radiation: 1.4Gy for 5 days to the liver metastasis before chemoimmunotherapy. Chemoimmunotherapy: gemcitabine(1000mg per square meter on days 1,8) , cisplatin (80mg per square meter on day 1), penpulimab (200mg, day1)

SUMMARY:
This study aims to evaluate the efficacy and toxicity of adding low-dose radiotherapy to chemoimmunotherapy as a first-line treatment for nasopharyngeal carcinoma patients with liver metastasis.

DETAILED DESCRIPTION:
Low-dose radiotherapy to the liver metastasis. Chemotherapy: gemcitabine and cisplatin Immunotherapy: penpulimab

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 70 years, male or non-pregnant female.
2. Histologically confirmed with nonkeratinizing carcinoma of the nasopharynx (differentiated or undifferentiated type, WHO II or III)
3. Stage IVB (AJCC 8th edition staging)
4. De novo nasopharyngeal carcinoma with liver metastasis, or patients who had received curative treatment (radical radiotherapy or radical radiotherapy combined with chemotherapy) and developed liver metastasis more than 6 months after treatment completion.
5. ECOG performance status: 0 or 1
6. Must have at least one measurable lesion (assessed according to RECIST v1.1)
7. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelets ≥ 100 × 10^9/L; hemoglobin ≥ 90 g/L.
8. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × upper limit of normal (ULN); activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
9. Serum creatinine ≤ 1.5 × ULN or estimated glomerular filtration rate (eGFR) ≥ 60 mL/min.
10. Serum total bilirubin ≤ 1.5 × ULN (patients with Gilbert's syndrome may be included if total bilirubin < 3 × ULN); AST and ALT ≤ 5 × ULN （because of liver metastasis）

Exclusion Criteria:

1. Patients with tumor recurrence at the primary site who have previously received radical radiotherapy.
2. Tumor invasion involving major blood vessels, with a high risk of significant bleeding as assessed by the investigator.
3. Systemic anticancer therapy, including hormone therapy, administered within 28 days prior to the initiation of the study treatment.
4. Previous treatment with immune checkpoint inhibitors (e.g., PD-1/PD-L1, CTLA-4).
5. Patients with active autoimmune diseases or a history of autoimmune diseases with a risk of recurrence.
6. Known history of other malignancies (except cured basal cell carcinoma or carcinoma in situ of the cervix).
7. Conditions requiring systemic corticosteroid therapy (equivalent to >10 mg/day of prednisone or similar medications) or other immunosuppressive therapy within ≤14 days prior to treatment.
8. Uncontrolled diabetes or laboratory abnormalities ≥Grade 1 in potassium, sodium, or corrected calcium levels despite standard treatment, or ≥Grade 3 hypoalbuminemia within ≤14 days before treatment.
9. History of the following diseases: interstitial lung disease, non-infectious pneumonitis, or uncontrolled diseases, including pulmonary fibrosis or acute lung disease.
10. Severe chronic or active infections requiring systemic antibiotics, antifungals, or antivirals within ≤14 days before the first dose of the investigational drug (including tuberculosis infection).
11. Known history of HIV infection.
12. Untreated chronic hepatitis B patients or hepatitis B virus (HBV) carriers with HBV DNA ≥500 IU/mL, or active hepatitis C virus (HCV) carriers.
13. Any major surgery requiring general anesthesia within ≤28 days prior to treatment.
14. Previous allogeneic stem cell transplantation or organ transplantation.
15. Any cardiovascular risk factors, including: cardiac chest pain that restricts daily instrumental activities ≤28 days before treatment. Symptomatic pulmonary embolism within ≤3 months before treatment. Acute myocardial infarction within ≤6 months before treatment. History of heart failure meeting New York Heart Association (NYHA) Class III or IV within ≤6 months before treatment. Grade ≥2 ventricular arrhythmias within ≤6 months before treatment. History of cerebrovascular accident within ≤6 months before the first dose of the investigational drug.
16. Evident bleeding tendencies or clinically significant bleeding symptoms ≤28 days prior to randomization, including but not limited to gastrointestinal bleeding, nasal bleeding (excluding epistaxis or retrograde blood-stained nasal discharge), and persistent bleeding disorders or coagulopathy.
17. Known allergy to any component of the investigational drug or a history of severe hypersensitivity to other monoclonal antibodies.
18. Peripheral neuropathy of Grade ≥2 as defined by NCI CTCAE v5.0.
19. Administration of live vaccines within ≤4 weeks prior to treatment.
20. Underlying medical conditions (including laboratory abnormalities) or alcohol/drug abuse or dependency that could impair drug administration, interpretation of drug toxicity, or adverse events (AEs), or could compromise study compliance or execution.
21. Pregnant or breastfeeding women.
22. Other factors deemed by the investigator that could lead to the premature termination of the study, such as other severe illnesses, significant laboratory abnormalities, or family/social factors that could affect participant safety or the collection of study data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Intrahepatic progression-free survival (iPFS) | 1 year
  Defined as the time from the start of therapy to the first progression in liver

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  Defined as the time from the start of therapy to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.
Overall survival (OS) | 2 year
  Defined as the time from the start of therapy to death from any cause or censored at the date of last follow-up.
Objective response rate (ORR) | 18 weeks
  Defined as the proportion of patients achieving complete response (CR) or partial response (PR) in all patients. According to RECIST 1.1 evaluation criteria, physicians use the efficacy evaluation record as the determination criteria
Incidence rate of adverse events (AEs) | 2 year
  Analysis of acute and late adverse events (AEs) are evaluated by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Qingnan Tang, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Huai Liu, Changsha, Hunan
  - Hui Wang, Changsha, Hunan
  - Qiyuan Zhou, Chenzhou, Hunan
  - Xinfu Liu, Shaoyang, Hunan
  - Jie Weng, Yueyang, Hunan

IPD SHARING:
Plan to Share IPD: No
Because of the policy of hospital